CLINICAL TRIAL: NCT05423327
Title: Cross-Sectional Study to Determine Distribution of Genetic Variants Among Subjects at Risk of, or With Known Non-alcoholic Steatohepatitis (NASH)
Brief Title: Genetic Data Collection in Adult Participants to Identify Genetic Variants of Known Importance in Non-alcoholic Steatohepatitis (NASH)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: R0000-NASH-CES-2117
Record Dates: First submitted 2022-06-01; First posted 2022-06-21 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Non-alcoholic Steatohepatitis (NASH)
Keywords: Nonalcoholic fatty liver disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: N/A: No study drug administered
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Blood Draw (Other)
  Interventions: Procedure: No Intervention

INTERVENTIONS:
Procedure: No Intervention — Single blood draw

SUMMARY:
Collection of clinical and genetic data to help identify individuals that carry genetic variants of known importance in Non-alcoholic Steatohepatitis (NASH)

ELIGIBILITY:
Key Inclusion Criteria:

One or more of the following:

1. A prior diagnosis of NASH with a Clinical Research Network (CRN) fibrosis score of F1 to F4 based on liver biopsy
2. Evidence of NAFLD by imaging or liver histology as described in the protocol

   * The possible imaging modalities to assess historic evidence of NAFLD may be based on thresholds as described in the protocol
3. Known high-risk genotype for HSD17B13 (T/T or T/TA) and/or PNPLA3 (C/G,or G/G)
4. A clinical suspicion of NASH based on presence of 2 or more elements of the metabolic syndrome defined by:

   1. Waistline that measures >35 inches (89 centimeters) for women or >40 inches (102 centimeters) for men
   2. Historic fasting triglycerides >150 mg/dL within the prior 6 months
   3. Historic fasting HDL cholesterol <40 mg/dL in men or <50 mg/dL in women, or on cholesterol-lowering medication within the prior 6 months
   4. Historic fasting blood glucose >100 mg/dL or on diabetes medication within the prior 6 months
   5. Historic blood pressure >130/85 mmHg, or on anti-hypertensive medication within the prior 6 months

Key Exclusion Criteria:

1. Known history or clinical evidence of drug abuse, within the 12 months before screening. Drug abuse is defined as compulsive, repetitive, and/or chronic use of drugs or other substances with problems related to their use and/or where stopping or a reduction in dose will lead to withdrawal symptoms.
2. Excessive alcohol intake for ≥3 months during the past year prior to screening (>3 units/day for males and >2 units/day for females is generally considered excessive (unit: 1 glass of wine [approximately 125 mL]=1 measure of spirits [approximately 1 fluid ounce]=½ pint of beer [approximately 284 mL]).
3. History of liver transplant, current placement on a liver transplant list, or Model for End-stage Liver Disease (MELD) score >12.
4. History of viral and resolved hepatitis or human immunodeficiency virus (HIV).
5. Any malignancy within the past 5 years except for basal cell or squamous epithelial cell carcinoma of the skin, or any carcinoma in situ.

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5311 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Genotype frequencies of rs72613567 in Hydroxysteroid 17β dehydrogenase 13 (HSD17B13) | Day 1
Genotype frequencies of rs738409 in patatin-like phospholipase domain containing 3 (PNPLA3) | Day 1

SECONDARY OUTCOMES:
Distribution of fibrosis-4 (FIB-4) scores across participants with different genotypes of rs72613567 in HSD17B13 | Day 1
Distribution of FIB-4 scores across participants with different genotypes of rs738409 in PNPLA3B13 | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (50):
- United States (30):
  - Southern California Research Center, Coronado, California
  - Velocity Clinical Research, Gardena, California
  - UCSD Health System, La Jolla, California
  - National Research Institute, Los Angeles, California
  - Clinnova Research Solutions, Orange, California
  - National Research Institute, Panorama City, California
  - FEMZ Clinical Research, Redondo Beach, California
  - Inland Empire Liver Foundation, Rialto, California
  - Precision Research Institute, Llc, San Diego, California
  - San Fernando Valley Health Institute, West Hills, California
  - Integrity Clinical Research, LLC, Doral, Florida
  - Miami Clinical Research, Miami, Florida
  - Genoma Research Group, Inc., Miami, Florida
  - US Associates in Research, LLC, Miami, Florida
  - Links Clinical Trials, Miami, Florida
  - Med Research Of Florida, LLC, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - IMIC, Inc, Palmetto Bay, Florida
  - Revival Research, Palmetto Bay, Florida
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - Mercy Medical Center, Inc, Baltimore, Maryland
  - University of Pennsylvania - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Mt. Olympus Medical Research, Friendswood, Texas
  - Mt. Olympus Medical Research, Houston, Texas
  - Synergy Group US LLC, Houston, Texas
  - Pioneer Research Solutions, Inc, Houston, Texas
  - Liver Center of Texas, Plano, Texas
  - Epic Medical Research, Red Oak, Texas
  - American Research Corporation at The Texas Liver Institute, San Antonio, Texas
  - R & H Clinical Research, Stafford, Texas
- Brazil (5):
  - Centro de Diabetes de Curitiba Ltda, Curitiba, Paraná
  - Hospital de Clínicas de Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul Ltda, Porto Alegre, Rio Grande do Sul
  - IBPClin-Instituto Brasil de Pesquisa Clínica - CCBR, Rio de Janeiro
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
- Mexico (5):
  - Grupo Médico Terranova - Hospital Terranova, Guadalajara, Jalisco
  - CEDOPEC - Centro Especializado en Diabetes, Obesidad y Prevención de Enfermedades Cardiovasculares, S.C., Miguel Hidalgo, Mexico City
  - PCR, Cuautitlán Izcalli, State of Mexico
  - Unidad de Atención Médica e Investigación en Salud (UNAMIS), Mérida, Yucatán
  - Investigación en Salud y Metabolismo S.C / Nutrición Clínica, Chihuahua City
- Puerto Rico (5):
  - Dr. Federico Rodriguez-Perez MD, Office of, San Juan
  - Latin Clinical Trial Center, San Juan
  - VA Caribbean Healthcare System, San Juan
  - Fundación de Investigación de Diego, Inc., San Juan
  - Dr. Paola Mansilla-Letelier MD, Office of, San Juan
- South Korea (5):
  - Keimyung University Dongsan Hospital, Dalseo-gu, Daegu
  - Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Hanyang University Seoul Hospital, Seoul, Gyeonggi-do
  - Chung-Ang University Hospital, Dongjak-gu, Seoul
  - Seoul National University Hospital, Jongno-gu, Seoul